CLINICAL TRIAL: NCT01808469
Title: A Randomized, Double Blind, Placebo-controlled, Pharmacokinetics/Pharmacodynamics-guided, Phase I Study in Healthy Volunteers Given Escalating, Single Intravenous Doses of NI-0101 in the Absence and Then in the Presence of a Systemic Lipopolysaccharide Challenge.
Brief Title: First in Human Study of an Anti-Toll-like Receptor 4 (TLR4) Monoclonal Antibody (NI-0101) in Adult Healthy Volunteers
Acronym: NI-0101-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Light Chain Bioscience - Novimmune SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NI-0101-01_
Record Dates: First submitted 2013-02-18; First posted 2013-03-11 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Antibodies, Monoclonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NI-0101 (Experimental): NI-0101 is an anti-Toll-like receptor monoclonal antibody.
  Interventions: Biological: Monoclonal antibody
- Placebo (Placebo Comparator): The placebo to be used for the proposed clinical trial is a sterile solution for intravenous infusion. The placebo is identical to the NI-0101 drug product but does not include the active substance.
  Interventions: Biological: Monoclonal antibody

INTERVENTIONS:
Biological: Monoclonal antibody

SUMMARY:
The purpose of this study is to determine the safety, tolerability and distribution and elimination of a novel therapeutic drug when administered to Healthy Volunteers. In addition its effects on some inflammatory parameters will be measured in presence or absence of lipopolysaccharide stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between 18 and 40 years old (inclusive) having a body mass index (BMI) between 18 and 30 kg/m2 (inclusive), able to adhere to study protocol requirements and having signed informed consent.

Exclusion Criteria:

* Any abnormal past or present clinically relevant medical history or any relevant abnormal laboratory parameters at screening that will prevent to consider the volunteers as healthy for the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of NI-0101 in healthy male/female subjects | Up to 8 weeks
  * 12 lead ECG
  * Vital signs
  * Physical examination
  * Adverse events
  * Routine laboratory assessments
  during 8 weeks post administration.

SECONDARY OUTCOMES:
Pharmacokinetic parameters of NI-0101 | Up to 8 weeks
  Blood samples for plasma NI-0101 concentrations.
  The following pharmacokinetic parameters of NI-0101 will be measured:
  Area under the curve from the time of dosing extrapolated to infinity (AUCinf); Area under curve from the time of dosing to the last measurable concentration (AUClast); AUCinf - AUClast expressed in % of AUCinf (% AUCextr); Systemic drug clearance (CL); Mean residence time (MRT) extrapolated to infinity (MRTinf); Mean residence time (MRT) at last measurable concentration (MRTlast).
Pharmacodynamic parameters of NI-0101 | Up to 8 weeks
  Blood samples for inflammatory markers measured in blood with or without the presence of an exogenous stimulus (lipopolysaccharide).
  Cytokine levels induced by ex vivo lipopolysaccharide challenge and circulating cytokine levels induced by in vivo lipopolysaccharide challenge will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: J. Koos Prof. Burggraaf, MD, Ph, Principal Investigator — Centre for Human Drug Research, Leiden, The Netherlands
Locations (1):
- Centre for Human Drug Research, Leiden, Netherlands